CLINICAL TRIAL: NCT05283954
Title: Use of a Combined Regimen of Fluoxetine, Prednisolone and Ivermectin in the Treatment of Mild COVID-19 to Prevent Disease Progression in Papua New Guinea: a Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Use of a Combined Regimen of Fluoxetine, Prednisolone and Ivermectin in the Treatment of Mild COVID-19 to Prevent Disease Progression Progression in Papua New Guinea
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Oriol Mitja (Other)
Collaborators: National Department of Health, Papua New Guinea (Unknown); Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor-Investigator, Oriol Mitja, Community Health Program Director, Lihir Medical Centre
Organization: Lihir Medical Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fluo-Pred-Iver
Record Dates: First submitted 2022-03-16; First posted 2022-03-17 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: SARS-CoV2 Infection; COVID-19
Keywords: Ivermectin; Fluoxetin; Prednisolone
MeSH Terms: conditions — COVID-19 | interventions — Prednisolone; Ivermectin; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined Regime of Fluoxetine, Prednisolone and Ivermectin (Experimental): Fluoxetine: 20mg tablet; 20 mg; once daily for 10 days; oral
  Prednisolone: 25 mg tablet; 25mg; once daily for 5 days; oral
  Ivermectin: 3 mg tablet; 0.4 mg/kg; once daily for 5 days; oral
  Interventions: Drug: Combination regimen: Fluoxetine, Prednisolone, Ivermectin
- Combination of Vitamin C and Albendazole (Other): Vitamin C: 50 mg tablet; 1 tablet; Once daily for 10 days; Oral
  Albendazole; 200 mg; 1 tablet; Once daily for 5 days; Oral
  Vitamin C: 50 mg tablet; 0.13 tablet/kg*; Once daily for 5 days; Oral
  *Same number of tablets than for Ivermectin
  Interventions: Drug: Combination regimen: Albendazole, Vitamin C

INTERVENTIONS:
Drug: Combination regimen: Fluoxetine, Prednisolone, Ivermectin — Subjects will receive the following treatments:
  Fluoxetine 20 mg oral tablets: One tablet right after randomization (Day 0) followed by one daily tablet for the following 09 days.
  Prednisolone 25 mg oral tablets: One tablet right after randomization (Day 0) followed by one daily tablet for the following 04 days.
  Ivermectin 3 mg oral tablets: Tablets started right after randomization (Day 0; 400mcg/ kg dosing), administered once a day for 05 consecutive days.
  Arms: Combined Regime of Fluoxetine, Prednisolone and Ivermectin
Drug: Combination regimen: Albendazole, Vitamin C — Subjects will receive the following treatments:
  Vitamin C 50 mg oral tablets: One tablet right after randomization (Day 0) followed by one daily tablet for the following 09 days.
  Albendazole 200 mg oral tablets: One tablet right after randomization (Day 0) followed by one daily tablet for the following 04 days.
  Vitamin C 50 mg oral tablets: Tablets started right after randomization (Day 0; 130mcg/ kg dosing), administered once a day for 05 consecutive days.
  Arms: Combination of Vitamin C and Albendazole

SUMMARY:
The Fluo-Pred-Iver clinical trial will test the efficacy of a combined regimen of Fluoxetine, Prednisolone and Ivermectin (Fluo-Pred-Iver), as treatment for ambulatory patients with mild COVID-19. The overarching idea of the work proposed herein is to investigate the use of Fluo-Pred-Iver to treat COVID-19, conducting a randomized controlled clinical trial to evaluate a new indication for these widely available drugs. It is estimated to include 954 participants.

DETAILED DESCRIPTION:
In this study, individuals who have a confirmed SARS-CoV-2 infection, as determined by a PCR or antigen rapid diagnostic test within the last 5 days, will be informed about the study.

Interested participants will be screened for eligibility criteria by research study staff. After review of inclusion and exclusion criteria, informed consent will be obtained. Participants who consent will be randomized to receive a combined regimen of Fluoxetine, Prednisolone and Ivermectin (Fluo-Pred-Iver), or a combined regimen of Albendazole and Vitamin C as control.

Patients will be followed remotely and/or in persona with visits on day 3, 7, 10 and 14 after inclusion. The primary objective will be to measure the proportion of a composite endpoint of moderate, severe or critical COVID-19 (as defined by NIH) and Emergency Department attendance of hospitalization, or death up to day 14. The reduction of SARS-CoV-2 viral load at day 7 measured by RT-qPCR will also be evaluated.

As secondary endpoints, the therapeutic potential of early administration of the combined regimen Fluo-Pred-Iver in reducing WHO Clinical progression scale score and the safety and tolerability of Fluo-Pred-Iver will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female individuals of ≥18 years old.
2. In women of childbearing potential, negative pregnancy test at inclusion/baseline visit.
3. Has confirmed SARS-CoV-2 infection as determined by PCR, a validated NAAT (i.e., GeneXpert), or validated antigen rapid diagnostic test from nasopharyngeal swabs ≤5 days prior to inclusion/baseline visit.
4. Symptomatic with mild COVID-19 with symptoms onset date ≤ 7 days prior to inclusion/baseline visit. Mild COVID-19, as defined per NIH: Individuals who have any of the common signs and/or symptoms of COVID-19 (i.e., fever, cough, sore throat, malaise, headache, muscle pain) without shortness of breath, dyspnoea, or abnormal chest imaging.
5. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
6. Has understood the information provided and capable of giving informed consent.

Exclusion Criteria:

1. If female, pregnant or breastfeeding, or planning a pregnancy during the study.
2. Moderate COVID-19, as defined per NIH:

   a. Moderate COVID-19: Individuals who have evidence of lower respiratory disease by clinical assessment or imaging and a saturation of oxygen (SpO2) ≥94% on room air at sea level.
3. Severe or critical COVID-19, as defined per NIH:

   1. Severe COVID-19: respiratory frequency >30 breaths per minute, SpO2 <94% on room air at sea level, ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300 mmHg, or lung infiltrates >50%.
   2. Critical COVID-19: respiratory failure, septic shock, and/or multiple organ dysfunction.
4. History of previous confirmed SARS-CoV-2 infection.
5. History of significantly abnormal liver function (Child Pugh C).
6. History of chronic kidney disease (CKD) ≥ stage 4 or need of dialysis treatment.
7. Any pre-existing condition that increases risk of thrombosis.
8. History of allergic reactions to ivermectin, fluoxetine, prednisolone, or vitamins C, albendazole, any of its excipients.
9. Concomitant use of medications that are highly dependent of CYP 2D6 for clearance and for which elevated plasma concentrations may be associated with serious and/or life-threatening events.

   1. Phenytoin
   2. Tricyclic antidepressants
   3. Antipsychotics: phenothiazines (i.e., chlorpromazine) haloperidol and most atypical (i.e., amitriptyline, aripiprazole, brexpiprazole, risperidone).
   4. Donepezil
   5. Tamoxifen
   6. Antiarrhytmics: propafenone, flecainide
   7. Amphetamine
10. Concomitant use of SSRIs, SNRIs, or tricyclic antidepressants, linezolid, or methylene blue (rationale: increased risk of serotonin syndrome or TCA overdose).
11. Concomitant use of drugs that could prolong the QT interval:

    1. Specific antipsychotics: ziprasidone, iloperidone, chlorpromazine, mesoridazine, droperidol
    2. Specific antibiotics: erythromycin, gatifloxacin, moxifloxacin, sparfloxacin
    3. Class 1A antiarrhytmics: amiodarone, sotalol
12. Concomitant use of donepezil (S1R agonist) or sertraline (S1R antagonist)
13. Uncontrolled psychiatric disorders, or suicidal ideation.
14. Inability to consent and/or comply with study protocol, in the opinion of the investigator.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
COVID-19 disease progression | Up to 14 days after administration of investigational medicinal product (IMP)
  This is a composite endpoint of moderate, severe or critical COVID-19 and Emergency Room attendace or hospitalization, or death
SARS-CoV-2 viral load | Up to 7 days after administration of IMP
  Reduction in SARS-CoV-2 viral load in nasopharyngeal swabs at day 7 after start of treatment, as determined by RT-qPCR

SECONDARY OUTCOMES:
COVID-19 WHO Clinical progression scale score | Up to 14 days after administration of IMP
  Change in COVID-19 WHO Clinical progression scale score
Adverse Events | Up to 14 days after administration of IMP
  Incidence of Adverse Events